CLINICAL TRIAL: NCT00268749
Title: Glycine Treatment of Prodromal Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02T-175
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Glycine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: glycine

INTERVENTIONS:
Drug: glycine — 0.8 g/kg/day

SUMMARY:
This is an open label trial of the NMDA agonist glycine used alone for symptoms that appear to be prodromal for schizophrenia in adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

* age 14-35
* meets SIPS criteria for psychosis prodrome

Exclusion Criteria:

* current antipsychotic medication
* more than 4 weeks of antipsychotic medication lifetime

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2002-07; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Scale Of Prodromal Symptoms total score | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Woods, MD, Principal Investigator — Yale University

REFERENCES:
- [Derived] Woods SW, Walsh BC, Hawkins KA, Miller TJ, Saksa JR, D'Souza DC, Pearlson GD, Javitt DC, McGlashan TH, Krystal JH. Glycine treatment of the risk syndrome for psychosis: report of two pilot studies. Eur Neuropsychopharmacol. 2013 Aug;23(8):931-40. doi: 10.1016/j.euroneuro.2012.09.008. Epub 2012 Oct 22. PMID 23089076